CLINICAL TRIAL: NCT05090189
Title: The Influence of Exercise Training on Musculoskeletal Health in Patients With Systemic Lupus Erythematosus Who Undergo Glucocorticoid Pulse Therapy
Brief Title: Exercise and Nutrition Recommendations for Patients Using Glucocorticoids (ENRG)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bruno Gualano (Other)
Responsible Party: Sponsor-Investigator, Bruno Gualano, Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The ENRG Study
Record Dates: First submitted 2021-09-10; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: exercise; autoimmune; training; glucocorticoids
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study comprises a 6-month parallel-group, randomized, controlled trial, in which individuals with Systemic Lupus Erythematosus who have undergone glucocorticoid pulse therapy (500-1000mg/d methylprednisolone i.v., 1-3 days), will be randomized into one of two conditions: control, consisting of no intervention and standard medical care; and exercise training, consisting of standard medical care supplemented by a twice-weekly, home-based, remotely monitored exercise training program. Patients will be assessed at three timepoints, namely 1-3 weeks after pulse therapy (according to patient's health state and willingness, PRE); three months after baseline (MID); and six months after baseline (POST).
Masking Description: Given that this is an exercise trial, blinding of study participants or investigators is not possible. Whenever possible, outcome assessors (e.g., lab technicians) will be blinded to the participants allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): The experimental arm will enroll in a 6-month, twice-weekly, home-based, remotely monitored exercise training program, the emphasis of which will be to improve musculoskeletal health and function.
  Interventions: Other: Exercise Training
- Control (No Intervention): The control group will receive standard medical care.

INTERVENTIONS:
Other: Exercise Training — The present intervention will consist of a 6-month long, twice-weekly, home-based, monitored exercise training program, with training sessions lasting around 40 minutes, with 48 sessions in total. The program will be delivered in the form of 6 x 4-week "blocks", which will progressively increase in intensity and complexity, as the participants physical capacities develop. Additionally, and in addition with current physical activity guidelines, participants will be instructed to perform at least an additional 70 minutes of purposeful activities per week. Study trainers will discuss the content of these activities with each individual participant to facilitate selection of suitable activities (e.g., brisk walking, jogging, stair climbing or bike riding), but their selection will be left to the discretion of the individual participants, and activity logs will be maintained throughout the study period.
  Arms: Exercise training

SUMMARY:
This parallel-group randomized, controlled, clinical trial aims to investigate the influence of a 6-month home-based, remotely-monitored, exercise training intervention on musculoskeletal health in patients with Systemic Lupus Erythematosus who have undergone glucocorticoid pulse therapy.

DETAILED DESCRIPTION:
Glucocorticoid treatment is a frequently prescribed to individuals with autoimmune diseases, such as Systemic Lupus Erythematosus, due to its anti-inflammatory effects. This treatment strategy has proven clinical benefits, but it can also adversely influence musculoskeletal health. Glucocorticoid pulse therapy is a particularly intensive treatment strategy, commonly used when the disease state is at its most active. Patients who undergo pulse therapy have a high risk of muscle and bone loss, and exercise training is a promising adjunct therapy to potentially ameliorate these adverse effects, but the feasibility and efficacy of this approach has yet to be investigated. The aim of this study, therefore, is to conduct a parallel-group, controlled, randomized clinical trial, to investigate the feasibility and efficacy of a home-based, remotely-monitored, exercise training intervention on musculoskeletal health in patients with Systemic Lupus Erythematosus who have undergone glucocorticoid pulse therapy.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 18 to 45 diagnosed with Systemic Lupus Erythematosus according to SLICC criteria;
* Medical indication and prescription for glucocorticoid pulse therapy;
* Access to Internet and any device that allows for participation in exercise training online lessons (such as smart phone, laptop or personal computer);
* Willingness to participate in an exercise training program.

Exclusion Criteria:

* Any physical, mental, neurological or musculoskeletal health impairment that contra-indicates exercise training.
* Use of medical therapy that alters bone metabolism, such as bisphosphonates, teriparatide and denosumab;
* Receiving prescription for multiple glucocorticoid pulse therapies mid-intervention;
* Being currently enrolled or having enrolled in a structured exercise training program in the last 6 months (defined as at least 2 planned, structures sessions of exercise training per week);
* Having a vertebral fracture at the moment of enrollment (identified by Vertical Fracture Assessment), or high risk for fracture (defined as low hip or spine bone mass [z-score < -3] or history of fragility fractures).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Bone health | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by dual-energy X-ray absorptiometry, high resolution peripheral quantitative computed tomography and blood bone biomarkers (C-terminal telopeptide [β-CTX-1], procollagen type 1 amino-terminal propeptide [P1NP], sclerostin, osteocalcin).

SECONDARY OUTCOMES:
Muscle health | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by dual-energy X-ray absorptiometry (fat-free mass), one-repetition maximum test (bench press and leg extension), and muscle functionality tests (timed-up-and-go, timed-stands, handgrip).
Aerobic capacity | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by maximal graded ergospirometric test.
Body composition | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by dual-energy X-ray absorptiometry (fat mass, percentage body fat, lean mass), body mass index, waist and hip circumferences.
Intervention feasibility and acceptability | Entire study duration.
  Assessed by feasibility metrics: Recruitment Capacity, Acceptability and Suitability, Resources, and Intervention Efficacy.
Cardiovascular risk | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by Framingham Risk Score
Proinflammatory cytokines | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by interferon gamma (IFN-γ), interleukin 10 and 6 (IL-10, IL-6), tumor necrosis factor alpha (TNF-α), and soluble TNF receptors (sTNFR1 e sTNFR2) assays.
Nutritional intake | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by three non-consecutive food recalls.
Disease activity | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K).
General quality of life | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  36-Item Short Form Survey (SF-36).
Disease-related quality of life | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by Systemic Lupus Erythematosus Quality of Life Questionnaire (SLEQOL)
Physical activity levels | Baseline (PRE), after 3 months (MID), and after 6 months (POST).
  Assessed by International Physical Activity Questionnaire (IPAQ)
Current and past bone-loading physical activity levels | Baseline (PRE).
  Assessed by Bone-Specific Physical Activity Questionnaire (BPAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Eimear Dolan, PhD, Principal Investigator — Faculdade de Medicina FMUSP, Universidade de Sao Paulo, Sao Paulo, SP, BR
Locations (1):
- Clinical Hospital of the School of Medicine, University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
On study completion, and once data has been analysed and submitted for publication, anonymised individual participant data for all outcomes will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: Anonymised data will be made permanently available upon study completion and once data has been analysed and submitted for publication.
Access Criteria: Anonymised data will be accessible to anyone interested via online repositories.